CLINICAL TRIAL: NCT02424929
Title: Asleep Versus Awake Deep Brain Stimulation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1994
Record Dates: First submitted 2015-04-14; First posted 2015-04-23 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2017-04

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Masking Description: Randomized parallel assignment, unblinded
Oversight: Data Monitoring Committee: No

ARMS (2):
- Awake (Other): Original surgery intervention.
  Patient will have DBS surgery done in the normal fashion. Asleep for the drilling of the burr holes, then awakened for the placement of the electrodes. No intervention will be given.
  Interventions: Procedure: Original Surgery
- Asleep (Other): Sedation intervention.
  Surgical intervention, anesthesia will be administered during entire placement of the system. Patient will not be awake at any point during procedure. All other aspects of surgery will be conducted normally.
  Interventions: Procedure: Sedation

INTERVENTIONS:
Procedure: Sedation — Propofol anesthesia administered during entire surgery.
  Arms: Asleep
Procedure: Original Surgery — No intervention, surgery will be conducted as usual. With sedation only during the drilling of the burr holes.
  Arms: Awake

SUMMARY:
The goal of this study is to compare the surgical outcome of deep brain stimulation (DBS) surgery in patients who are deeply sedated, "asleep," or not sedated, "awake," during surgical implantation of the DBS electrode. The investigators hypothesize that the clinical outcome, neurophysiological findings, and surgical accuracy will be equivalent. There are 3 specific aims: 1) compare the activity of the neurons in the patients' brain in the asleep and awake groups using microelectrode recording, to see how this affects clinical outcome capability of microelectrode recordings and macrostimulation to identify the subthalamic nucleus in asleep patients. 2) Determine if intraoperative CT scans of the DBS electrode is sufficient for accurate DBS electrode placement. 3) Compare the clinical outcome on their Parkinson's disease between awake and asleep DBS patients.

DETAILED DESCRIPTION:
All patients will undergo DBS surgery using regular surgical techniques. In this surgery a halo is attached to the skull. A CT scan is obtained. MRI - based targeting is conducted to identify to target location to implant the electrode deep in the brain. The patients have a burr hole placed just behind their hair line in the frontal lobe. Then a guide tube is inserted in the brain. Neurophysiological identification and confirmation of the target is conducted with multiple techniques including microelectrode recording to listen to single neurons in the brain, and macrostimulation to test clinical effect. The electrode is implanted and its clinical effect is tested. The halo is removed and the patient is taken to the recovery room. Patients will be randomized to undergo the surgery awake or asleep. Our current standard surgical technique is awake with intravenous anesthesia used briefly during drilling of a burr hole in the skull.

But in selected cases patients have remained sedated throughout the entire surgery. Patients in the asleep group will have intravenous anesthesia maintained throughout the entire case.

Standard intraoperative neurophysiological and imaging techniques will be used. In awake patients these techniques are used to identify and confirm that the DBS electrode is implanted in accurate position. These techniques include microelectrode recording where individual neurons are monitored as the electrode is inserted through the brain tissue. Early research reports suggest that sedation may affect the neuronal activity. But our preliminary data indicates that is still reliable under intravenous anesthesia. Macrostimulation using the implanted DBS electrode can suppress tremor, stiffness, and slowness of Parkinson's disease, and assists in confirmation of electrode position. It also causes side effects including tingling, and facial contractions. These methods will also be studied in the asleep patients. The O-arm is an intraoperative CT scanner that visualizes the DBS electrode. O-arm images will be obtained in the standard fashion in both groups. The accuracy of intraoperative imaging will be compared to standard postoperative MRI. The clinical outcome from these two techniques will be compared. The clinical outcome will be measured with standard Parkinson's disease research tools including video taped and independently rated motor exam, as well as the Unified Parkinson's Disease Rating Scale (UPDRS). Gait analysis will be collected using the APDM system. These will be tested before and at 3 months after surgery by the neurologist.

ELIGIBILITY:
Inclusion Criteria:

* All patients will have moderate to advanced Parkinson's disease.
* Patients must be medically safe for asleep or awake surgery.
* Ability to speak English well.

Exclusion Criteria:

* Parkinson's patients with concurrent dementia as measured by neurocognitive testing, or with significant strokes identified on MRI will be excluded. Other similar diseases will be excluded from the study such as Essential Tremor, and Parkinson's plus disorders.
* Patients that are obese or that have severe potential airway issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2025-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Lead Placement | 6 months post operation
  Determination of location of lead placement and efficacy of programming. x,y,z coordinates related to the anterior commissure and posterior commissure.

SECONDARY OUTCOMES:
Stimulation Parameters | 6 months post operation
  Record stimulation settings. Contacts, voltage, frequency, pulse width.
Unified Parkinson's Disease Rating Scale-UPDRS | 1 month pre-operation and 6 month post operation
  Compare UPDRS score pre and post surgery
Medication Data | 1 month pre-operation and 6 month post operation
  Compare medication dosage pre and post surgery; mg per dose, dose frequency, total dose, L-dopa equivalent.
Operation Data | Day of operation
  Microelectrode recordings Anesthesia record; anesthesia dose in reference to Ramsay Scale Stimulation side effects; where parasthesias are present (arm, leg, face), tremor, eye deviation, rigidity, hand speed.
Mobiltiy Lab | 1 month pre-operation and 6 month post operation
  Gait evaluation; jerkiness, time-domain (m/s^2, Hz), Frequency, temporal gait, cadence, stride length, range of motion, asymmetry, turning time, number of steps, anticipatory postural amplitude, duration.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Carlson, M.D Ph.D., Principal Investigator — Inland Neurosurgery and Spine
Locations (1):
- Providence Inland Neurosurgery & Spine, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes